CLINICAL TRIAL: NCT06778421
Title: Pilot Study to Identify the Impact of OnabotulinumtoxinA (BOTOX®) on Patient Perceived Stress.
Brief Title: Impact of OnabotulinumtoxinA (BOTOX®) on Stress
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Center for Advanced Facial Plastic Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTIIT-955A
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Stress (Psychology); Stress; Healthy Adult Female Participants; Stress, Psychologic; Stress, Psychological Cumulative; Stress, Physiological; Stress Response; Stress Levels; Stress Perception
Keywords: stress; BOTOX; PSS; Perceived stress scale; injection; reduction; BTA; facial rejuvenation; aesthetic procedure; psychological impact; clinical trial; facial expressions; stress relief; stress reduction; chemodenervation
MeSH Terms: conditions — Stress, Psychological; Fractures, Stress; Facial Expression | interventions — Injections, Intramuscular; Botulinum Toxins, Type A; Injections; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline (Placebo Comparator): Sterile, preservative-free 0.9% Sodium Chloride Injection, United States Pharmacopeia (USP) Only
  Interventions: Procedure: Intramuscular injection; Other: Sodium Chloride
- OnabotulinumtoxinA (BOTOX®) injection (Experimental): Active drug reconstituted with sterile, preservative-free 0.9% Sodium Chloride Injection, United States Pharmacopeia (USP) Only
  Interventions: Procedure: Intramuscular injection; Drug: OnabotulinumtoxinA (Botox®) Injections

INTERVENTIONS:
Procedure: Intramuscular injection — Injection performed using method for aesthetic facial rejuvenation procedure with neuromuscular chemodenervation agents
Drug: OnabotulinumtoxinA (Botox®) Injections — Injection of 64 units of active drug at a ratio of 4 units to 0.1 mL of sterile, preservative-free 0.9% Sodium Chloride Injection, United States Pharmacopeia (USP) Only
  - Abbvie/Allergan drug.
  Other Names: Botulinum Toxin A; BTA
  Arms: OnabotulinumtoxinA (BOTOX®) injection
Other: Sodium Chloride — Placebo injection of the same volume of preservative-free 0.9% Sodium Chloride Injection, United States Pharmacopeia (USP) Only.
  Arms: Saline

SUMMARY:
The purpose of this prospective single-center, blinded*, randomized, proof-of-concept study is to determine whether OnabotulinumtoxinA (BOTOX®) injections will change the level of stress perceived by generally healthy adult female participants. It is hypothesized that BOTOX® injections will be associated with decreases in perceived stress levels, measured by scores on the Perceived Stress Scale (PSS) questionnaire. The primary outcome measure is a chronological decrease in PSS scores between any two points of the study period.

Comparison of the placebo- and BOTOX®-treated participant scores will either support or disprove the study hypothesis.

Qualified participants who meet the study requirements, including a one-time completion of basic laboratory testing before treatment.

The treatment visit starts on day-1 of a 12-week period, which consists a total of four clinic visits and one online visit, which involve:

* vital signs and Body Mass Index (BMI) measurements
* basic/interval history and physical
* 2 Perceived Stress Scale (PSS) questionnaires
* injection of 64 units of either BOTOX® or sterile salt solution
* stay for 60-minutes after treatment for monitoring and to complete study tasks

DETAILED DESCRIPTION:
Note: The initial phase of this study is limited to those who are assigned female sex at birth, for reasons of treatment dosing only. This study does not have any gender-specific requirements. Future, larger studies, if indicated, will likely be open to all participants.

* Intervention type is masked for both the participant and the treating physician. However, this is subject to change in the case of adverse reactions or events.

Please contact study affiliates for additional information.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects capable of giving informed consent in the English language
2. Females 18-65 years of age
3. Perceived Stress Scale (PSS) ≥ 14 at screening.
4. Participants who have been toxin-naive for ≥1 year (i.e. onabotulinumtoxinA (BOTOX®), alternatives, or its derivatives)
5. Female subjects willing to minimize the risk of inducing pregnancy for the duration of clinical study
6. Subjects in good physical and mental health and not on any prescription psychiatric medications
7. Subjects willing to not undergo any other aesthetic or skin treatments for the duration of the study

Exclusion Criteria:

1. Participants with history of facial (including periorbital) surgery within the last 12 months
2. Use of neuromodulators in the past ≤ 12 months
3. History or known alcohol and/or illicit drug abuse
4. Participants with psychiatric diagnosis
5. Body Mass Index (BMI) at Screening ≥ 30 kg/m2.
6. Participants with metabolic disorders (e.g., hypothyroidism and hyperparathyroidism)
7. Undiagnosed, unstable, or preexisting conditions that in the opinion of the investigators, would interfere with the course and conduct of the study. These include but are not limited to inflammatory disorders, diseases that affect muscles and/or nerves such as myasthenia gravis and Lambert-Eaton syndrome, high blood pressure, heart disease, and/or stroke that could result in a life-threatening response when treated with BOTOX® or placebo.
8. Participant has any laboratory abnormality (found on screening) that, in the opinion of the investigators, is clinically significant, has not resolved at baseline and could jeopardize or would compromise the participant's ability to participate in this study.
9. Prior use of isotretinoin
10. Active skin disease or infection at or near injection sites
11. Active use of tobacco or nicotine products in any form via any route (e.g. inhalation, ingestion, absorption)
12. Chronic marijuana or tetrahydrocannabinol exposure
13. If the investigators feel that the subject is not a good candidate for the study
14. Females of childbearing potential not using a reliable means of contraception
15. Female subjects must not be breastfeeding
16. Any known previous hypersensitivity reactions to BOTOX®
17. Current or recent (within therapeutic window) use of neuromuscular medications that may pose additional risk with treatment with BOTOX®, such as but not limited to amino-glycosides and anticholinergic drugs

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Changes in Perceived Stress Scale (PSS) | within 12-13 weeks of intervention
  Chronological decrease at any two points between the first and last completed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Babak Azizzadeh, MD, FACS, Principal Investigator — Center for Advanced Facial Plastic Surgery; Marielle He, MD, MS, Principal Investigator — Center for Advanced Facial Plastic Surgery
Locations (1):
- Center for Advanced Facial Plastic Surgery, Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Time frame of study-related information availability and duration is dependent on study progression and the actual date of completion. This will be updated promptly when the investigators are able to provide an estimate of the projected end-date.
Access Criteria: TBD.
  Access criteria are currently under development and infrastructure is not yet established. The criteria will be available upon finalization of these processes and regulatory and stakeholder review and approval.